CLINICAL TRIAL: NCT02243995
Title: Physical Training in Sarcoidosis Patients With Fatigue Complaints
Brief Title: Physical Training in Sarcoidosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ild care foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC 12-3-032
Record Dates: First submitted 2013-02-18; First posted 2014-09-18 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2014-09

CONDITIONS: Sarcoidosis
Keywords: Training program; Resistance training; Endurance training; Muscle strength; Exercise capacity; Fatigue; Quality of life
MeSH Terms: conditions — Sarcoidosis; Fatigue | interventions — Physical Conditioning, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Physical training (Experimental)
  Interventions: Other: Physical training; Behavioral: Physical training

INTERVENTIONS:
Other: Physical training
Behavioral: Physical training

SUMMARY:
Exercise intolerance, muscle weakness and fatigue complaints are frequent and persistent problems in sarcoidosis. These physical impairments are disabling and affect quality of life in a negative way. The aetiology of these physical impairments is multifactorial. Physical inactivity can cause deconditioning, resulting in more perceived fatigue and muscle weakness. These symptoms may be partially reversible following a structured physical training program. However, scientific studies about physical training in sarcoidosis are lacking. Therefore, the aim of the present study is to examine the changes in fatigue complaints, physical functioning and quality of life (QOL) in patients with sarcoidosis following a 13-week physical training program.

After obtaining written informed consent, sarcoidosis patients will start a 13-week physical training program for three times a week. This training program includes peripheral muscle training for both the upper and lower extremities (starting at 40% of the multiple-repetition maximum) and endurance training consisting of walking on a treadmill (starting at 60% of the speed of the 6-minute walk test) or cycling on a ergometer (starting at 50% of the Wmax).

Participants will be assessed at baseline (week 0), at the end (13 weeks) and 3 months after ending the training. During these assessments, patients perform muscle strength (m. quadriceps and m. biceps) and exercise tests (six-minute walk test and submaximal endurance cycling test). They also complete several questionnaires:

Fatigue Assessment Scale (FAS), World Health Organization Quality of Life assessment instrument-BREF (WHOQOL-BREF), Small Fiber Neuropathy Screening List (SFNSL), Medical Research Council (MRC), Visual Analogue Scale (VAS) and Hospital Anxiety and Depression Scale (HADS)

ELIGIBILITY:
Inclusion Criteria:

* Patients are diagnosed with sarcoidosis according to the WASOG guideline.
* Fatigued patients ((FAS-score ≥ 22 points) and/or a reduced six-minute walking distance (predicted six-minute walking distance -50 m).
* Patients who signed the consent form and are able to participate in a training program.
* Minimum age 18 years and maximum age 70 years.
* Clinically stable: no exacerbation of complaints, or changes in initiated therapeutic management during the preceding 3 months.

Exclusion Criteria:

* Patients with a cognitive failure, making them unable to understand questionnaires and instructions.
* Patients with a oncological, cardiac, neurological or orthopedic history making them unable to participate in a training program.
* Patients who are unfamiliar with the Dutch language, disabling them to understand questionnaires and instructions.
* Patients who participated in a physical training program six months prior to inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Cange in Fatigue Assessment Scale (FAS)at 3 months after end of the training | baseline (week 0), at the end (week 13) and 3 months after ending the training
  The 10-item FAS is a fatigue scale. Each item has a 5-point rating scale and FAS scores range from 10-50. FAS scores <22 indicate nonfatigue persons and scores of 22-34 indicate fatigued persons.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine F. Lenssen, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Fysiomedica, Geleen, Limburg, Netherlands

REFERENCES:
- [Background] Marcellis RG, Lenssen AF, de Vries GJ, Baughman RP, van der Grinten CP, Verschakelen JA, De Vries J, Drent M. Is there an added value of cardiopulmonary exercise testing in sarcoidosis patients? Lung. 2013 Feb;191(1):43-52. doi: 10.1007/s00408-012-9432-6. Epub 2012 Nov 9. PMID 23138855
- [Background] Marcellis RG, Lenssen AF, Elfferich MD, De Vries J, Kassim S, Foerster K, Drent M. Exercise capacity, muscle strength and fatigue in sarcoidosis. Eur Respir J. 2011 Sep;38(3):628-34. doi: 10.1183/09031936.00117710. Epub 2011 Mar 24. PMID 21436356
- [Derived] Marcellis R, Van der Veeke M, Mesters I, Drent M, De Bie R, De Vries G, Lenssen A. Does physical training reduce fatigue in sarcoidosis? Sarcoidosis Vasc Diffuse Lung Dis. 2015 Jun 22;32(1):53-62. PMID 26237356
- See also: ild care foundation — http://ildcare.eu